CLINICAL TRIAL: NCT04983446
Title: A Phase 2 Proof-of-concept Study to Evaluate the Safety, Tolerability, and Efficacy of Intranasal Foralumab in Hospitalized Subjects With Severe COVID-19 and Pulmonary Inflammation
Brief Title: In-patient COVID-19 Study of Intranasal Foralumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to business reasons
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TILS-016
Record Dates: First submitted 2021-07-14; First posted 2021-07-30 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Covid19; COVID-19 Lower Respiratory Infection; COVID-19 Respiratory Infection
MeSH Terms: conditions — COVID-19 | interventions — foralumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to receive intranasal foralumab 100 µg (50 µg in 0.1 ml solution into each nostril) or placebo (0.1 ml vehicle solution into each nostril).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a Phase 2, randomized, placebo-controlled, double-blind, proof-of-concept study of intranasal foralumab in hospitalized subjects with severe COVID-19 and pulmonary inflammation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foralumab Arm + Standard of Care (Experimental): Subjects in this arm would receive, intranasal foralumab 100 µg (50 µg in 0.1 ml solution into each nostril).
  Interventions: Drug: Foralumab
- Placebo Arm + Standard of Care (Active Comparator): Subjects in this arm would receive, placebo (0.1 ml vehicle solution into each nostril).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Foralumab — Foralumab is a second generation fully human anti-CD3 antibody
  Arms: Foralumab Arm + Standard of Care
Other: Placebo — Placebo will be the vehicle for the foralumab nasal solution without active drug (25 mM sodium acetate/125 mM sodium chloride/0.02% polysorbate 80, pH 5.5 buffer).
  Arms: Placebo Arm + Standard of Care

SUMMARY:
This is a Phase 2, randomized, placebo-controlled, double-blind, proof-of-concept study of intranasal foralumab in hospitalized subjects with severe COVID-19 and pulmonary inflammation.

Foralumab is a fully human second generation anti-CD3 mAb with a modified Fc unit (two amino acid substitutions) composed of 2 heavy chains with an immunoglobulin (Ig) G1constant region and 2 light chains with a kappa constant region.

In a separate Phase 2 randomized, controlled, pilot trial conducted to assess safety, tolerability, and efficacy in 39 patients with mild to moderate COVID-19 in Brazil, showed that intranasal foralumab may be of benefit in modulating immune reactivity and in reducing pulmonary inflammation. Importantly, intranasal administration of foralumab was well tolerated with no clinically significant changes in blood cell counts (including blood lymphocytes), no evidence of hypersensitivity, and no serious adverse events (SAEs) were reported in the study.

DETAILED DESCRIPTION:
Approximately 80 hospitalized subjects with severe COVID-19 and evidence of pulmonary involvement on a computed tomography (CT) scan at screening will be enrolled in this study over 4 months, depending on enrollment. Up to 7 centers in Brazil will conduct this study.

The main study objective is to evaluate the effect of intranasal foralumab on evolution of pulmonary infiltrates in hospitalized subjects with severe COVID-19 pneumonia.

Subjects will be randomized 1:1 to receive intranasal foralumab 100 µg (50 µg in 0.1 ml solution into each nostril) or placebo (0.1 ml vehicle solution into each nostril). All subjects will receive continued Standard of Care (SoC) therapy (per hospital/study site policies and guidelines) together with intranasal foralumab or placebo for the entire 14-day treatment period.

Subjects will participate in the study approximately 35 days (from screening to completion).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age hospitalized with severe COVID-19, who are within 2 weeks of symptom onset.
2. Laboratory-confirmed SARS-CoV-2 infection as determined by nucleic acid amplification test (NAAT) from an upper respiratory specimen within 72 hours of randomization. Test type and result must be documented in the study record.
3. Subject agrees to the collection and processing of blood and saliva samples, non-invasive oxygen monitoring (via pulse oximeter), nasal speculum examination, and radiography (high-resolution CT scanning) as required in the protocol.
4. Subject (or their legally authorized representative [LAR]) is willing and able to provide written informed consent.
5. Has at least 2 of the following symptoms for ≥ 48 hours: fever or history of fever (oral temp ≥ 38°C), cough, headache, fatigue, muscle aches, gastrointestinal symptoms, and/or shortness of breath.
6. Respiratory rate ≥ 30 per minute, SpO2 ≤ 93% on room air at sea level, heart rate ≥ 125/min, and/or PaO2/FiO2 < 300.
7. Radiologic evidence of pneumonia (infiltrates on high-resolution CT) at screening.
8. Erythrocyte sedimentation rate (ESR), CRP and/or lactate dehydrogenase (LDH) > upper limit of normal [ULN] at screening.

Exclusion Criteria:

1. Age < 18 years.
2. Subject has a body mass index >35 kg/m2 or glycosylated hemoglobin (Hgb A1c) ≥ 9% at screening.
3. Currently requires (or in opinion of Investigator is likely to require within 48 hours of enrollment) mechanical ventilation or extracorporeal membrane oxygen saturation (ECMO).
4. Prior history (or considered to be at risk) of acute liver disease or chronic unstable liver disease (Child-Pugh B or C) OR alanine transaminase (ALT) or aspartate transaminase (AST) > 5 × ULN at screening.
5. Prior history of chronic obstructive pulmonary disease requiring supplemental oxygen, or active/incompletely treated tuberculosis.
6. Concomitant uncontrolled systemic bacterial or fungal infection OR concomitant viral infection other than COVID-19 (e.g., Influenza, respiratory syncytial virus).
7. Any underlying condition or therapy associated with immunosuppression.
8. Serious concomitant illness which in the opinion of the Investigator precludes the subject from enrolling in the trial.
9. History of untreated syphilis, hepatitis B, or untreated hepatitis C virus.
10. Uncontrolled human immunodeficiency virus.
11. Acute kidney injury Stage 3 or higher or chronic kidney disease Stage 4 or higher.
12. Known hypersensitivity to foralumab or excipients.
13. Females of child-bearing potential, who are pregnant, breast-feeding, intend to become pregnant or are not using highly effective contraceptive methods. Females who are postmenopausal (defined as at least 12 months of amenorrhea) are not considered to be of child-bearing potential. Highly effective contraceptive methods are defined as:

    1. Having a male partner who is sterile (vasectomized or orchiectomized) prior to the female subject's entry into the trial and is the sole sexual partner for that female subject
    2. Surgically sterile (hysterectomy or bilateral oophorectomy); bilateral tubal ligation with surgery at least 6 weeks before study initiation
    3. Use of intra-uterine devices in place for at least 3 months
    4. Stable hormonal contraception for at least 3 months before study initiation and through study completion
    5. Barrier method (condom or diaphragm) with spermicide for at least 14 days before study initiation through study completion
    6. True abstinence: When this is in line with the preferred and usual lifestyle of the subject (period abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
14. Active participation in any other clinical trial or receipt of an experimental treatment within the preceding 30 days.
15. Receipt of COVID-19 convalescent plasma, or COVID-19 mAbs, within 3 months of enrollment.
16. Receipt of any anti-IL-6 mAb or similar anti-inflammatory medications (e.g, Janus kinase inhibitors) within 3 months of enrollment.
17. Prior receipt of any COVID-19 vaccine.
18. Receipt of any treatment for COVID-19 (off-label, compassionate use, or investigational use) except per local SoC within 30 days prior to screening.
19. History of opioid or cocaine (including crack cocaine) use.
20. Use of any nasally administered medications within 1 week of enrollment.
21. In the opinion of the Investigator, the subject is unable to comply with the requirements to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of intranasal foralumab on evolution of pulmonary infiltrates in hospitalized subjects with severe COVID-19 pneumonia | Day 14 and Day 28
  It is determined based on change from baseline in semiquantitative chest CT severity score.A chest CT severity score was calculated by assessing the degree of lobe involvement for each of the five lung lobes separately as follows: 0% (no involvement), 1%-25% (minimal involvement), 26%-50% (mild involvement), 51%-75% (moderate involvement), and 76%-100% (severe involvement). Higher the score the worse the outcome.

SECONDARY OUTCOMES:
To evaluate the effect of intranasal foralumab on resolution of severe COVID-19 as assessed by chest CT severity score | Day 14 and Day 28
  Proportion of randomized subjects with chest CT severity score < 19.5
To evaluate the safety of intranasal foralumab when administered up to 14 days | Day 28
  Adverse events categorized and graded via CTCAE
To assess the impact of intranasal foralumab on nasal symptoms when administered up to 14 days | Day 14
  Change from baseline in subject-reported Intranasal Tolerability Rating Scale (ITRS). ITRS is rated on an 11-point scale, ranging from 0 (none) to 10 (worst I can imagine) and consists of 3 questions.

IPD SHARING:
Plan to Share IPD: No